CLINICAL TRIAL: NCT07382765
Title: In This toGether: Testing a Population-based Text Messaging-based HIV Prevention Program for Young Adults Across Uganda
Brief Title: In This toGether R01
Acronym: ITG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Makerere University (Other); Internet Solutions for Kids Uganda (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH136955 (NIH); R01MH136955 (NIH)
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: HIV
MeSH Terms: interventions — Film Dosimetry

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention)
- Quiz and badge (Experimental): Receives quiz and badge interactive elements
  Interventions: Other: Level up quizzes; Other: Badges; Other: Content
- Bagde and buddy (Experimental): Badges and advice are the only interactive elements
  Interventions: Other: Badges; Other: On-demand advice; Other: Content
- Quiz and buddy (Experimental): Advice buddy and level up quizzes are only interactive parts of intervention
  Interventions: Other: Level up quizzes; Other: On-demand advice; Other: Content
- No interactive elements (Experimental): Receives educational content with no interactive elements
  Interventions: Other: Content

INTERVENTIONS:
Other: Level up quizzes — Participant is given weekly quiz questions on that week's texted content
  Arms: Quiz and badge; Quiz and buddy
Other: Badges — Participants can earn badges by performing activities encouraged by program
  Arms: Bagde and buddy; Quiz and badge
Other: On-demand advice — Participants have access to ITGenie/Text Buddy, which responds to keywords with preset messages
  Arms: Bagde and buddy; Quiz and buddy
Other: Content — Texted information about HIV prevention
  Arms: Bagde and buddy; No interactive elements; Quiz and badge; Quiz and buddy

SUMMARY:
The goal of this study is to assess the effectiveness of the text-based ITG intervention to promote behaviors associated with HIV prevention amongst 18-22 year-olds in Uganda.

The main questions the study aims to answer are:

1. In a twelve-month period, does the intervention increase HIV testing and use of condoms?

   a. How do the different interactive elements effect this?
2. How is effectiveness different for populations based on education, sex, and location (urban/rural)? Researchers will compare the control group, with no intervention, and the three combinations of the three intervention components: quiz questions, milestone badges, and access to on-demand advice.

Participants will receive the intervention via text messages and partake in the interactive elements listed above.

ELIGIBILITY:
Inclusion Criteria:

* Live in Uganda
* Age 18 to 22
* Have exclusive ownership of a cell phone
* Have used text messaging for at least 6 months
* Able to read English, Luganda, Runyakitara, or Luo

Exclusion Criteria:

* Not participated in preliminary R34 study

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
HIV testing | 12 months
  Binary variable. Was the participant tested for HIV during the study?
Condom-protected sex acts | 12 months
  Self-reported count of condom-protected sex acts during study

CONTACTS AND LOCATIONS:
Locations (1):
- Internet Solutions for Kids Uganda, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collins LM, Kugler KC, Gwadz MV. Optimization of Multicomponent Behavioral and Biobehavioral Interventions for the Prevention and Treatment of HIV/AIDS. AIDS Behav. 2016 Jan;20 Suppl 1(0 1):S197-214. doi: 10.1007/s10461-015-1145-4. PMID 26238037
- [Background] Leddy MJ. Spirit that matters. CHAC Rev. 1996 Summer;24(2):8-11. No abstract available. PMID 10159628
- [Background] Matovu J, Wanynze R, Kasozi D. Assessment of the implementation processes and outcomes of the HIV assisted partner notification program in Uganda. Kampala: Makerere University School of Public Health. Published online July 2021.
- [Background] Bogart LM, Musoke W, Mukama CS, Allupo S, Klein DJ, Sejjemba A, Mwima S, Kadama H, Mulebeke R, Pandey R, Wagner Z, Mukasa B, Wanyenze RK. Enhanced Oral Pre-exposure Prophylaxis (PrEP) Implementation for Ugandan Fisherfolk: Pilot Intervention Outcomes. AIDS Behav. 2024 Oct;28(10):3512-3524. doi: 10.1007/s10461-024-04432-w. Epub 2024 Jul 19. PMID 39028385